CLINICAL TRIAL: NCT04270916
Title: Identifying the Prevalence, Severity and the Impact on Quality of Life of Long-term Ototoxicity in Cancer Survivors: a Cross-sectional Study
Brief Title: Prevalence and Impact on QoL From Ototoxicity in Cancer Survivors
Status: Suspended | Type: Observational
Why Stopped: due to COVID-19
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); International Stem Cell Forum (Other)
Responsible Party: Sponsor
Other Study IDs: 19039
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hearing Loss, Sensorineural; Tinnitus, Subjective; Cancer; Chemotherapeutic Toxicity
MeSH Terms: conditions — Hearing Loss, Sensorineural; Tinnitus; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High frequency pure tone audiometry — Hearing test carried out routinely, non invasive

SUMMARY:
This study will involve collaborating with oncologists in the post-chemotherapy follow-up appointments. The participants who wish to consent to this study will then answer 3 short questionnaires (THI, HHIA and SF-36) about hearing loss, tinnitus and quality of life. The audiologist or the researcher, under the supervision of an audiologist, will then perform a simple, non-invasive hearing test on the participant. Should the participant have a hearing loss, they will be advise to seek help from their General Practitioner.

DETAILED DESCRIPTION:
There has been a substantial increase in cancer survival rates in the the past decades, however many cancer survivors are now impacted by the multitude of toxicities associated with treatment. It is only when temporary toxicities subside that the long-term toxicities progress and become important. Chemotherapy, although highly effective, is known to cause ototoxicity, presenting as hearing loss and tinnitus. Hearing loss and tinnitus are associated with a higher risk of depression, dementia, social isolation and anxiety. There is little information and support offered to patients who suffer from ototoxicity, which can potentially lead to many being undiagnosed and untreated. Ototoxicity can be permanent and progressive, therefore it is essential that a deeper understanding and increased awareness of how hearing loss and tinnitus affects the quality of life (QoL) of cancer survivors can improve long-term symptoms Management and support offered.

This project aims to identify the prevalence and severity of long-term ototoxicity in cancer survivors following platinum-based treatment. Prevalence of ototoxicity can be unreliable and varies in the medical literature, with studies reporting rates between 24% and 79%. Information on prevalence will be achieved by recruiting patients from oncology clinics and performing a high frequency audiogram. The results from the audiogram will be compared to an normative dataset in addition to detecting self-reported hearing loss from the Hearing Handicap Inventory for Adults (HHIA) and the Hearing Handicap Inventory for Elderly (HHIE) questionnaires. Furthermore, the severity and prevalence of tinnitus will also be detected by using the Tinnitus Handicap Inventory (THI) questionnaire. A validated questionnaire assessing QoL (SF-36) after cancer will also be completed by the patients. The questionnaires will be statistically analysed and compared against a dataset from the general population in the hope to identify the concerns surrounding long-term ototoxicity in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent

  * Age 18+ at time of cancer diagnosis
  * At least 1 cycle of any type of platinum-based chemotherapy
  * 0-5 years following first cycle of platinum-based chemotherapy
  * Comprehensive understanding of the English language

Exclusion Criteria:

* Previous radiotherapy to the head and neck area
* Pre-existing hearing deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to identify the prevalence of hearing loss and tinnitus and the impact on quality of life in people who have been treated with platinum based chemotherapy anywhere from 0-5 years ago. They can have any type of cancer as long as they were adults at the time of diagnosis and were treated with cisplatin, carboplatin or oxaliplatin.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire | Afer 6 months
  Short form 36 item questionnaire to assess quality of life (0-100 scale, higher score means better outcome)

SECONDARY OUTCOMES:
Hearing loss | After 6 months
  High frequency audiogram (PTA)
Hearing Handicap Inventory for adults/elderly | After 6 months
  Self reported hearing loss using the HHIA/HHIE questionnaire (0-100, higher score means more handicap)
Tinnitus Handicap Inventory | After 6 months
  Self reported tinnitus using the THI questionnaire (0-100 with higher scoring being more handicap)

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Personal data will not be shared, however the overall statistical results grouping the cohort will be.